CLINICAL TRIAL: NCT00209781
Title: Effect of Intermittent Preventive Treatment (IPTp) With Sulfadoxine-Pyrimethamine Plus Insecticide Treated Nets, Delivered Through Antenatal Clinics for the Prevention of Malaria in Mozambican Pregnant Women
Brief Title: IPTp Plus ITNs for Malaria Control in Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: TimNet
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Pregnancy
MeSH Terms: interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Sulfadoxine-Pyrimethamine (Fansidar)
Device: ITNs

SUMMARY:
We aim to evaluate whether IPT in pregnancy provides any additional benefit to the protection afforded by ITNs.

DETAILED DESCRIPTION:
Pregnant women are at an increased risk for malaria infection and disease. Maternal anaemia, low birth weight and prematurity are the most frequent adverse effects of the infection. The current WHO recommendation consists on the provision of insecticide treated nets (ITN's) and intermittent preventive treatment (IPT). Results from a recentn trial of ITN's have shown a significant reduction in maternal anaemia, parasitaemia and low birth weight prevalence in women sleeping under impregnated nets. However, scarce information exists on the relative efficacy of IPT and ITNs to reduce the deleterious effects of malaria infection during pregnancy when given at the same time. This information is of relevance to guide national malaria control programmes.

This study consists on the administration of two double blind doses of IPT with Sulfadoxine-Pyrimethamine or placebo at predefined intervals, after the beginning of the second trimester. All women receive an ITN.

ELIGIBILITY:
Inclusion Criteria:

* Less than 28 weeks of pregnancy

Exclusion Criteria:

* Previous allergic reactions to sulphonamides

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1028
Dates: Start 2003-08; Study Completion 2006-12

PRIMARY OUTCOMES:
Evaluate whether two doses of intermittent treatment with SP delivered through antenatal clinics provides additional benefit to the protection afforded by ITNs on low birth weight

SECONDARY OUTCOMES:
To assess whether intermittent treatment with sulfadoxine-pyrimethamine provides any additional benefit to the protection afforded by ITNs on the:
Maternal anaemia at and after delivery
Parasite prevalence at and after delivery
Placental malaria infection
Infant mortality and morbidity
Gestational age of the newborn
Child parasitaemia and anaemia 12 months after delivery
To identify the operational and socio-cultural issues involved in the delivery to and use of ITNs by pregnant women
To evaluate the cost-effectiveness of the interventions
To determine the duration of the efficacy of long-lasting insecticide-treated nets against Anopheles mosquitoes
To assess the immunological protection against malaria in children during the first year of life regarding malaria preventive interventions in their mothers during pregnancy
To asses the effect of IPT with SP in HIV positive pregnant women on the prevention of mother-to-child HIV transmission and on the viral load reduction in the mother

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Principal Investigator — Centre for International Health, Hospital Clinic de Barcelona
Locations (1):
- Centro de Investigaçao em Saude da Manhiça, Manhiça, Maputo Province, Mozambique

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Mayor A, Moro L, Aguilar R, Bardaji A, Cistero P, Serra-Casas E, Sigauque B, Alonso PL, Ordi J, Menendez C. How hidden can malaria be in pregnant women? Diagnosis by microscopy, placental histology, polymerase chain reaction and detection of histidine-rich protein 2 in plasma. Clin Infect Dis. 2012 Jun;54(11):1561-8. doi: 10.1093/cid/cis236. Epub 2012 Mar 23. PMID 22447794
- [Derived] Bardaji A, Sigauque B, Sanz S, Maixenchs M, Ordi J, Aponte JJ, Mabunda S, Alonso PL, Menendez C. Impact of malaria at the end of pregnancy on infant mortality and morbidity. J Infect Dis. 2011 Mar 1;203(5):691-9. doi: 10.1093/infdis/jiq049. Epub 2011 Jan 3. PMID 21199881
- [Derived] Sicuri E, Bardaji A, Nhampossa T, Maixenchs M, Nhacolo A, Nhalungo D, Alonso PL, Menendez C. Cost-effectiveness of intermittent preventive treatment of malaria in pregnancy in southern Mozambique. PLoS One. 2010 Oct 15;5(10):e13407. doi: 10.1371/journal.pone.0013407. PMID 20976217
- [Derived] Menendez C, Bardaji A, Sigauque B, Sanz S, Aponte JJ, Mabunda S, Alonso PL. Malaria prevention with IPTp during pregnancy reduces neonatal mortality. PLoS One. 2010 Feb 26;5(2):e9438. doi: 10.1371/journal.pone.0009438. PMID 20195472
- [Derived] Serra-Casas E, Menendez C, Bardaji A, Quinto L, Dobano C, Sigauque B, Jimenez A, Mandomando I, Chauhan VS, Chitnis CE, Alonso PL, Mayor A. The effect of intermittent preventive treatment during pregnancy on malarial antibodies depends on HIV status and is not associated with poor delivery outcomes. J Infect Dis. 2010 Jan 1;201(1):123-31. doi: 10.1086/648595. PMID 19954383
- [Derived] Naniche D, Lahuerta M, Bardaji A, Sigauque B, Romagosa C, Berenguera A, Mandomando I, David C, Sanz S, Aponte J, Ordi J, Alonso P, Menendez C. Mother-to-child transmission of HIV-1: association with malaria prevention, anaemia and placental malaria. HIV Med. 2008 Oct;9(9):757-64. doi: 10.1111/j.1468-1293.2008.00626.x. Epub 2008 Jul 19. PMID 18651857
- [Derived] Menendez C, Bardaji A, Sigauque B, Romagosa C, Sanz S, Serra-Casas E, Macete E, Berenguera A, David C, Dobano C, Naniche D, Mayor A, Ordi J, Mandomando I, Aponte JJ, Mabunda S, Alonso PL. A randomized placebo-controlled trial of intermittent preventive treatment in pregnant women in the context of insecticide treated nets delivered through the antenatal clinic. PLoS One. 2008 Apr 9;3(4):e1934. doi: 10.1371/journal.pone.0001934. PMID 18398460
- See also: Related Info — http://www.manhica.org